CLINICAL TRIAL: NCT01119469
Title: Dysfunctional Illness-related Cognitions in Individuals With Hypochondriasis and Change Thereof
Brief Title: Comparing Cognitive Therapy and Exposure Therapy in Individuals With Hypochondriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Florian Weck, PhD, Goethe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WE 4654/2-1, WE 4654/2-3
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Hypochondriasis; Somatoform Disorders
Keywords: Hypochondriasis; Health Anxiety; randomized controlled trial; Cognitive Therapy; Exposure Therapy
MeSH Terms: conditions — Hypochondriasis; Somatoform Disorders | interventions — Psychotherapy; Cognitive Behavioral Therapy; Implosive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive Therapy (CT) (Experimental): There will be 12 50-minute individual sessions conducted at weekly intervals. Booster sessions will be conducted one, three and six months after treatment. Sessions include psychoeducation, attention training, cognitive restructuring, behavioral experiments, imagery rescripting and relapse prevention.
  Interventions: Behavioral: Psychotherapy (CT or ET)
- Exposure Therapy (ET) (Experimental): There will be 12 50-minute individual sessions conducted at weekly intervals. Booster sessions will be conducted one, three and six months after treatment. Sessions include change of safety behavior, exposition (in sensu and in vivo), and response prevention.
  Interventions: Behavioral: Psychotherapy (CT or ET)
- Waiting List (WL) (No Intervention): 12 weeks waiting time

INTERVENTIONS:
Behavioral: Psychotherapy (CT or ET) — weekly 50-minute sessions for 12 weeks
  Other Names: Cognitive Therapy; Exposure Therapy
  Arms: Cognitive Therapy (CT); Exposure Therapy (ET)

SUMMARY:
This study will compare the efficacy of cognitive therapy and exposure therapy for treating hypochondriasis.

DETAILED DESCRIPTION:
Hypochondriasis is defined as a preoccupation with the fear of having a serious disease based on the person's misinterpretation of bodily symptoms (APA). For a long time hypochondriasis was seen as difficult to treat. Meanwhile effective psychological treatment for hypochondriasis exists. Psychotherapies using cognitive therapy (CT), cognitive behavioral therapy (CBT), exposure therapy (ET) or behavioral stress management approaches are effective in reducing symptoms of hypochondriasis. However, few studies compare different types of psychotherapy. In addition, in these studies numbers of participants were small, no differences between different treatments were found, and one third of the participants showed no satisfactory change. This study will compare the efficacy of CT and ET in a larger sample of 84 participants.

Participants in this randomized controlled trial (RCT) will first undergo baseline assessment. Then they will be randomly assigned to either CT, ET or a waiting list (WL), all conditions are for the duration of 12 weeks. CT includes psychoeducation, attention training, cognitive restructuring, behavioral experiments, imagery rescripting and relapse prevention. ET includes change of safety behavior, exposition (in sensu and in vivo), and relapse prevention. Both treatment trials contain the identical number of sessions. Treatment response will be assessed at week 12 and additionally one and three years after treatment. Participants of the WL will be assigned to CT or ET after the waiting period.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for hypochondriasis
* German fluency and literacy
* Informed consent

Exclusion Criteria:

* Major medical illness expected to worsen significantly
* Currently in psychotherapy
* Suicidal tendency
* Clinical diagnosis of alcohol or drug addiction, schizophrenia, schizoaffective disorder or bipolar disorder according to DSM-IV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Hypochondriasis Yale-Brown Obsessive-Compulsive Scale (H-YBOCS) | 3 months
  clinician-rated measure that assesses hypochondriacal obsessions, compulsions and avoidance

SECONDARY OUTCOMES:
Illness Attitude Scales (IAS) | 3 months
  self-report measure that assesses attitudes, fears, and beliefs associated with the psychopathology of hypochondriasis and that of abnormal illness behavior
Beck-Depression Inventory II (BDI-II) | 3 months
  self-report measure that assesses depressive symptoms
Beck Anxiety Inventory (BAI) | 3 months
  self-report measure that asessses anxiety symptoms
Brief Symptom Inventory (BSI) | 3 months
  self-report measure that assesses aspects of general psychopathology
Scale for the Assessment of Illness Behavior (SAIB) | 3 months
  self-report measure that focuses on illness behavior
Health-related quality of life (SF-12) | 3 months
  self-report measure the assesses the health-related quality of life
Cognitions About Body and Health Questionnaire (CABAH) | 3 months
  self-rated measure that focuses on attitudes related to the cognitive concept of hypochondriasis

CONTACTS AND LOCATIONS:
Overall Officials: Florian Weck, PhD, Principal Investigator — Goethe University
Locations (1):
- Department of Clinical Psychology and Psychotherapy of the Wolfgang Goethe University, Frankfurt am Main, Hesse, Germany